CLINICAL TRIAL: NCT03799679
Title: Nanoparticle Albumin-Bound Paclitaxel Followed by Dose-Intensive Epirubicin in Combination With Cyclophosphamide as Neoadjuvant Chemotherapy in Triple Negative Breast Cancer
Brief Title: Albumin-Bound Paclitaxel Followed by Epirubicin in Combination With Cyclophosphamide in Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1808189-7
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Triple Negative Breast Cancer
Keywords: Neoadjuvant Chemotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Antineoplastic Agents

STUDY DESIGN:
Intervention Model Description: This is an open-label, single arm, two-stage Simon Design study for women with Triple Negative Breast Cancer. Patients will treated by Nanoparticle Albumin-Bound Paclitaxel Followed by Dose-Intensive Epirubicin in Combination with Cyclophosphamide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Experimental): Nanoparticle Albumin-Bound Paclitaxel 125mg/m2, iv, d1* 12 cycles ( weekly), followed by epirubicin 90mg/m2, iv, d1 + cyclophosphamide 600mg/m2, iv, d1 * 4 cycles (14 days per cycle)
  Interventions: Drug: Chemotherapeutic Agent

INTERVENTIONS:
Drug: Chemotherapeutic Agent — Drug: Nanoparticle Albumin-Bound Paclitaxel Nanoparticle Albumin-Bound Paclitaxel 125mg/m2, iv, d1. Patients will receive this as a single-agent for the first twelve weeks, then followed by epirubicin in combination with cyclophosphamide.
  Drug: Epirubicin 90 mg/m² given IV
  Drug: Cyclophosphamide 600 mg/m² given IV

SUMMARY:
This is an open-label, single arm, two-stage Simon Design study for women with Triple Negative Breast Cancer treated with Nanoparticle Albumin-Bound Paclitaxel and Carboplatin.

The primary objective of the trial is to evaluate of the efficacy and safety of weekly Nanoparticle Albumin-Bound Paclitaxel(Nab-P) Followed by Dose-Intensive Epirubicin in Combination with Cyclophosphamide as Neoadjuvant Chemotherapy in Triple Negative Breast Cancer.

The primary endpoint of the study is to to assess Pathological complete response rate（pCR）using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1)..

The total number of patients to be included in this study is 60 patients.

The duration of the study, from first patient visit to last patient visit will be approximately 19 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age: from 18 to 70 years old, female.
2. Has histologically or cytologically confirmed unilateral primary invasive breast cancer with a clinical stage of T2-4NanyM0.
3. The expression of ER, PR, HER-2 was negative by immunohistochemistry (IHC), if HER2 expression is 2+ patients need to be confirmed by in situ hybridization to detect no HER-2 gene amplification.
4. At least one measurable objective lesion according to RECIST 1.1 criteria.
5. ECOG performance status of 0-1.
6. LVEF≥55%.
7. Bone marrow function: Neutrophils ≥ 1.5×109/L, platelets ≥ 100×109/L, and hemoglobin ≥ 90 g/L.
8. Liver and renal function: Serum creatinine ≤ 1.5 times the upper limit of normal. AST and ALT ≤ 2.5 times the upper limit of normal Total bilirubin ≤ 1.5 times the upper limit of normal, or ≤ 2.5 times the upper limit of normal in patients with Gilbert's syndrome.
9. Has good compliance with the planned treatment, understand the study process and sign written informed consent.

Exclusion Criteria:

1. Any prior cytotoxic chemotherapy, endocrine therapy, biological therapy, or radiation therapy.
2. Patients with grade II or higher heart disease scored by the New York Heart Association (NYHA).
3. Severe systemic infection, or with other serious diseases.
4. Patients with known hypersensitivity or intolerance to chemotherapeutic agents or their excipients.
5. Other malignancies have occurred in the past 5 years, except for cured cervical carcinoma in situ, non-melanoma skin carcinoma.
6. Pregnant or lactating, and who refuse to take appropriate contraception during the course of this trial.
7. Have participated in other study studies within 30 days prior to the first dose of study drug.
8. Patients who, in the opinion of the Investigator, are not suitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is pathological complete remission (pCR) | 2 months
  Histopathological examination of breast and axillary lymph node specimens without invasive cancer cell remnants. Complete pathological response is also considered to be achieved if only in situ cancer cell remnants are present in the surgical specimens.

SECONDARY OUTCOMES:
The second endpoint includes the objective response rate (ORR) | 2 months
  The second endpoint ORR composed of tumor response classifications of complete response (CR) and partial response (PR), refers to the number of cases with complete and partial response after treatment as a percentage of the total number of evaluable cases.
Breast conserving surgery(BCS) rate | 2 months
  Percentage of patients undergoing breast-conserving surgery after neoadjuvant therapy as a whole evaluable.
Adverse events (AE) | 2 months
  Adverse events (AE) were monitored on an ongoing basis and classified according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03. Patients were assessed for toxicities before each administration, and toxicity was graded accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Principal Investigator — Fudan University
Locations (1):
- Cancer Hospital/ Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu Y, Fan L, Wang ZH, Shao ZM. Nab-paclitaxel Followed by Dose-dense Epirubicin/Cyclophosphamide in Neoadjuvant Chemotherapy for Triple-negative Breast Cancer: A Phase II Study. Oncologist. 2023 Jan 18;28(1):86-e76. doi: 10.1093/oncolo/oyac223. PMID 36426808